CLINICAL TRIAL: NCT07217756
Title: Influence of Body Mass Index on Gingival Health, White Spot Lesions, Whole Salivary Proinflammatory Cytokine and Adipokine Profile and Candida and Streptococcus Mutans Carriage Among Adolescents Undergoing Fixed Orthodontic Therapy
Brief Title: Impact of Increased Body Mass Index on Adolescent Fixed Orthodontic Treatment. A Prospective Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: American Association of Orthodontists Foundation (Unknown)
Responsible Party: Principal Investigator, Dimitrios Michelogiannakis, Associate Professor, Program Director of the Orthodontics Department, University of Rochester
Other Study IDs: STUDY00005905
Record Dates: First submitted 2025-10-15; First posted 2025-10-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obesity & Overweight; Orthodontic Treatment
Keywords: body mass index; obesity; orthodontic treatment; adolescents; fixed orthodontic appliances
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will collect and retain unstimulated whole salivary samples from the study participants. The investigators will also collect and retain gingival crevicular fluid samples, which will be collected with periopaper strips from the distal side of the six mandibular anterior teeth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Increased BMI group (test group): The increased BMI group will include patients with a BMI>25.0 Kg/m2.
- Normal BMI group (control groups): The normal-BMI group will include patients with a BMI between 18.5 and 24.99 (Kg/m2).

SUMMARY:
The goal of this prospective observational study is to assess the influence of increased body mass index (BMI) on various oral health and orthodontic-related parameters in adolescents undergoing orthodontic therapy (OT) with braces. These parameters include gum inflammation, tooth decalcifications/discolorations, tooth alignment of lower incisors, and various inflammatory and microbiological parameters in the collected saliva and gum fluid of the patients. The primary purpose is to assess if an increased BMI is a risk factor for oral inflammation in adolescents undergoing OT. The main questions it aims to answer are:

1. Do patients with an increased BMI undergoing OT demonstrate increased microbial counts in the saliva compared to patients with normal BMI?
2. Do patients with increased BMI undergoing OT demonstrate increased gum inflammation, tooth discolorations, and higher levels of inflammatory markers in the saliva and gum fluid samples compared to patients with normal BMI? This study will include 2 study groups (patients with increased BMI-test group, and normal weight patients-control group). The participants will be asked to complete a study questionnaire, which will collect information regarding their demographics, their family socioeconomic and educational status, dietary habits, and oral health-related quality of life. The participants will also receive an oral examination (evaluation of their gum health), and they will have their intraoral photos taken, as well as an impression of their lower teeth (to create dental models). A saliva sample will be obtained by asking patients to passively "drool" in a tube, and a gingival fluid sample will be collected from the gums of the lower anterior teeth using thin paper strips. All these study procedures will be conducted at baseline (T1: before bonding of braces), and at an approximately 6-month follow-up visit (T2). Comparisons of these outcomes will be conducted between the two groups and across timepoints.

ELIGIBILITY:
Inclusion Criteria:

* adolescents (12-17 years old);
* patients scheduled to undergo comprehensive fixed orthodontic therapy (OT) (for at least 6 months with metal braces/wires) on both dental arches;
* patients with increased BMI (≥25.0 Kg/m2) (test-Group);
* patients with normal BMI [18.5-24.99 (Kg/m2)] (control-Group);
* patients with all 6 mandibular anterior teeth present and mild-to-moderate mandibular crowding (<7.5 mm);
* patients and parents/guardians willing to provide signed assent/permission.

Exclusion Criteria:

* self-reported habitual tobacco product users;
* patients with self-reported medical diseases such as hepatic diseases, blood disorders, cardiovascular diseases, HIV, diabetes mellitus, and viral infections;
* patients with craniofacial syndromes and/or cleft lip and palate;
* pregnant and/or lactating females (by self/parent report);
* edentulous individuals;
* patients with active or a history of periodontitis;
* patients having undergone surgical and/or non-surgical periodontal therapy within the past 6 months;
* patients with physical and/or mental/cognitive disabilities who are decisionally-impaired and not able to consent/assent for themselves;
* patients who reported use of medications such as antibiotics, steroids (inhalers and/or pills), non-steroidal anti-inflammatory drugs, and antimicrobial mouth-rinses within the past 3 months or those who require prophylactic antibiotics prior to dental procedures;
* patients undergoing cancer therapy;
* underweight patients (BMI less than 18.5 Kg/m2);
* patients with oral mucosal lesions such as median rhomboid glossitis and lichen planus;
* patients with clinically visible carious teeth.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent patients undergoing fixed orthodontic therapy at the Eastman Institute for Oral Health, University of Rochester, NY.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Full-Mouth Bleeding Score (FMBS) | Baseline (T1: before bonding of braces) and approximately 6 months follow-up (T2)
  Bleeding on probing (BOP) will be assessed dichotomously (yes/no) at six sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual/palatal, mid-lingual/palatal, and disto-lingual/palatal) using a standardized periodontal probe by trained examiners. The full-mouth bleeding score (FMBS) will be calculated as the percentage of sites that bleed out of the total number of sites examined. Higher percentages indicate greater gingival inflammation.
Mean Change in White Spot Lesion (WSL) Score (International Caries Detection and Assessment System (ICDAS)) | Baseline (T1: before bonding of braces) and approximately 6 months follow-up (T2)
  Standardized intraoral and facial photographs will be taken using calibrated camera settings and stored in Dolphin Imaging Software. Each visible tooth surface will be examined for color, texture, and cavitation changes and scored using the International Caries Detection and Assessment System (ICDAS). Code 0 = sound surface; code 2 = visible white spot lesion; codes 3-4 = localized enamel breakdown or dentin shadowing; codes 5-6 = cavitated lesions extending into dentin. Because photos are obtained without air drying, code 1 will be excluded. The average WSL score per participant will be calculated by dividing the total ICDAS score by the number of surfaces assessed. Mean change = score at T2 minus score at T1. Higher scores indicate greater enamel decalcification.
Mean Change in Salivary Microbial Counts of Candida albicans and Streptococcus mutans | Baseline (T1: before bonding of braces) and approximately 6 months follow-up (T2)
  Unstimulated whole saliva will be collected at baseline and follow-up. C. albicans will be cultured on CHROMagar™ Candida and confirmed via germ tube test from three colonies per sample. S. mutans will be cultured on Mitis Salivarius Bacitracin medium and identified by colony morphology. DNA-based microbial identification and oral microbiome sequencing with bioinformatics analysis will also be performed. Microbial counts will be reported per participant as colony-forming units per milliliter (CFU/mL) or relative abundance. Higher values indicate greater microbial load.

SECONDARY OUTCOMES:
Mean Change in Body Mass Index (BMI) | Baseline (T1) and approximately 6 months follow-up (T2)
  Height (cm) will be measured using a stadiometer, and weight (kg) with a calibrated digital scale. BMI will be calculated as weight (kg)/height² (m²). Measurements will be taken twice and averaged. Higher BMI indicates greater body mass relative to height.
Mean Change in Full-Mouth Plaque Score (FMPS) | Baseline (T1) and approximately 6 months follow-up (T2)
  Plaque presence will be recorded on four surfaces per tooth (mesial, distal, buccal, lingual/palatal). The FMPS will be calculated as the percentage of surfaces with plaque present out of total surfaces examined. Higher percentages indicate poorer oral hygiene.
Mean Change in Percentage of Sites with Probing Depth >3 mm | Baseline (T1) and approximately 6 months follow-up (T2)
  Probing depth (PD) will be measured at six sites per tooth using a periodontal probe. The percentage of sites with PD greater than 3 mm will be calculated for each participant. Higher percentages indicate more severe periodontal disease.
Mean Change in Oral Dryness Score (Challacombe Scale) | Baseline (T1) and approximately 6 months follow-up (T2)
  Oral dryness will be assessed using the Challacombe Scale, which rates 10 indicators of xerostomia (e.g., lack of saliva pooling, frothy saliva, depapillation, fissured tongue). Scores range from 1 to 10, with 1-3 indicating mild dryness, 4-6 moderate, and 7-10 severe. Higher scores indicate greater dryness.
Mean Change in Little's Irregularity Index (Tooth Alignment) | Baseline (T1) and approximately 6 months follow-up (T2)
  Dental casts made from alginate impressions will be analyzed using a digital caliper (accuracy 0.01 mm). The sum of the linear displacements between the anatomic contact points of the mandibular incisors (five measurements) yields Little's Irregularity Index. Higher values indicate greater misalignment.
Mean Change in Salivary Proinflammatory Biomarker Concentrations (IL-1β, IL-6, TNF-α, Leptin, Resistin) | Baseline (T1) and approximately 6 months follow-up (T2)
  Salivary and gingival crevicular fluid samples will be centrifuged and analyzed using multiplexed magnetic bead assays (Milliplex MAP). Concentrations will be calculated from standard curves. Higher levels indicate greater inflammatory activity.
Mean Change in Dietary Habits Score | Baseline (T1) and approximately 6 months follow-up (T2)
  Participants will complete a standardized questionnaire assessing dietary habits related to oral health and obesity. Responses will be scored to produce a composite dietary habits score; higher scores indicate less healthy dietary patterns.
Mean Change in Oral Health-Related Quality of Life (OHIP-14 Total Score) | Baseline (T1) and approximately 6 months follow-up (T2)
  The Oral Health Impact Profile-14 (OHIP-14) questionnaire will assess functional limitation, pain, and psychological and social impacts of oral health. Scores from 14 items are summed (range 0-56); higher scores indicate poorer oral health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Michelogiannakis, DDS, MS, Principal Investigator — Eastman Institute for Oral Health, University of Rochester
Locations (1):
- Eastman Institute for Oral Health, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and the risk of re-identification, even with de-identified datasets. Additionally, the scope of consent obtained from participants during the trial does not include provisions for public sharing of individual-level data.